CLINICAL TRIAL: NCT02060617
Title: Impairment-Based Versus Classification-Based Physical Therapy for Acute and Subacute Low Back Pain: a Randomized Controlled Trial
Brief Title: A Comparison of Two Different Methods of Physical Therapy to Treat Acute and Subacute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hendricks Regional Health (Other)
Responsible Party: Principal Investigator, David Candy, Physical Therapist, Hendricks Regional Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-7
Record Dates: First submitted 2013-12-01; First posted 2014-02-12 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Low Back Pain
Keywords: low back pain; physical therapy; manual therapy; manipulation; exercise; motor control; regional interdependence
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impairment-Based Group (Experimental): The impairment-based intervention will be a multi-modal treatment approach utilizing manual therapy of the thoracolumbosacral spine and hips as well as motor control exercises. Patient education will also be provided.
  Interventions: Behavioral: Patient Education; Procedure: Manual therapy of the thoracolumbosacral spine and hips; Procedure: Motor control exercises
- Classification-Based Group (Active Comparator): Patients in this group will be categorized into subgroups according to the Treatment-Based Classification (TBC) Algorithm and treated accordingly. Patient education will also be provided.
  Interventions: Behavioral: Patient Education; Procedure: Treatment-Based Classification intervention

INTERVENTIONS:
Behavioral: Patient Education — All subjects will receive education that back pain is common but rarely harmful in nature, that pain does not necessarily mean that there is structural damage to their back, and that they should try to remain as active as they are able within the limits of their pain. In addition, individualized education regarding posture, body mechanics, sleeping positions, or other concerns of the patient will be provided on a pragmatic basis as deemed appropriate by the treating clinician.
Procedure: Manual therapy of the thoracolumbosacral spine and hips — Thrust and/or non-thrust manipulation and soft tissue mobilization as determined by mobility impairments identified on clinical examination.
  Arms: Impairment-Based Group
Procedure: Motor control exercises — Motor control exercises as determined by motor control impairments identified on clinical examination.
  Arms: Impairment-Based Group
Procedure: Treatment-Based Classification intervention — Lumbopelvic manipulation and range of motion exercise, spinal stabilization exercises, direction specific exercises, and/or traction will be applied as determined by the Treatment-Based Classification (TBC) Algorithm.
  Arms: Classification-Based Group

SUMMARY:
Recent research has shown that classifying patients with low back pain into treatment subgroups results in better improvements than treating all patients with low back pain the same. However, physical therapists may use different types of information to determine how to classify their patients. One method uses patient characteristics that have been shown by research to predict good results from a certain type of treatment. Another method uses specific impairments that the physical therapist identifies in a clinical exam to determine which treatment to provide. It is not currently known if one of these methods is better than the other. The purpose of this study is to determine if research-based classification or impairment-based treatment is more effective for treating patients with low back pain that has lasted less than 90 days in terms of improvements in pain and disability. The results of this study may help reduce the high financial cost associated with low back pain.

DETAILED DESCRIPTION:
PURPOSE: The purpose of this study is to describe a multimodal impairment-based clinical model for the treatment of low back pain utilizing the concept of Regional Interdependence (Wainner et al 2007) and to determine the relative effectiveness of this model versus classification-based therapy using the Treatment-Based Classification System for acute and subacute low back pain (Delitto et al 1995, Fritz et al 2006, Fritz et al 2007) in terms of improvements in pain and disability at 4 weeks and 6 months.

BACKGROUND: Recent studies have shown that subclassifying patients with low back pain into treatment groups results in better outcomes than treating all patients with low back pain as homogenous groups. (Fritz et al 2003) However, no studies have directly compared the efficacy of impairment-based versus classification-based physical therapy for patients with acute and subacute low back pain.

HYPOTHESIS: We suspect that both methods of treatment will be effective, but we are uncertain if one will be more effective than the other. Therefore, our null hypothesis will be that both methods will be equally effective.

METHODS:

1. Patients referred to physical therapy at Hendricks Regional Health in Plainfield, IN will be screened for eligibility. Eligible participants will be offered the opportunity to voluntarily participate in the research study. Those patients who are both eligible and interested will receive an informed consent form approved by the Hendricks Regional Health Institutional Review Board.
2. All subjects will complete a standard intake form and self-report measures. The principal investigator will obtain a subjective history from the patient and perform a standardized baseline physical examination.
3. After the baseline examination, subjects will be randomized in blocks of 4, 6, or 8 using a concealed, computer-generated randomization sequence accessed electronically through a Microsoft Excel spreadsheet using the VLOOKUP function to return the group assignment when the subject number is entered.
4. All subjects in both groups will be treated by the principal investigator two times per week for two weeks followed by once per week for two weeks (total of 6 visits) regardless of treatment group assignment. All subjects will receive standardized education as well as additional individualized education as deemed appropriate by the treating clinician. Subjects will be given a home exercise program consisting of the same exercises they performed in physical therapy and asked to perform their exercises twice per day.
5. Patients in the impairment-based group will be treated using a multi-modal treatment approach utilizing manual therapy of the thoracolumbosacral spine and hip as well as motor control exercises. Patients in the classification-based group will be categorized into subgroups according to the previously described Treatment-Based Classification (TBC) Algorithm and treated accordingly.
6. After completion of the 6 visits, we intend to discharge most patients to a home exercise program. However, patients who require more or fewer visits than this will still be included in the intention-to-treat analysis. Patients will be encouraged to perform their home exercises at least 3 times per week until the 6 month follow up.
7. Primary and secondary outcome measures will be collected at 4 weeks and 6 months from baseline.

DATA ANALYSIS:

Study data will be analyzed using SPSS Statistical Software (IBM, Armonk, NY).

1. Baseline characteristics will be examined for between group differences.
2. Primary outcomes will be analyzed using a repeated measures analysis of co-variance (ANCOVA) to examine a group x time interaction for pain and disability at baseline, 4 weeks, and 6 months controlling for baseline covariates of Fear Avoidance Behavior Questionnaire physical activity subscale score (FABQpa), duration of symptoms, and prior history of low back pain. Median and range values will be calculated for Global Rating of Change at 4 weeks and 6 month. Primary outcome measures will also be dichotomized and combined in order to determine overall treatment success for the 4 week and 6 month follow ups.
3. Intention-to-treat analysis using multiple imputation to account for missing values will be used in all analyses. A secondary per-protocol analysis will be performed for patients who completed exactly 6 visits, performed their home exercise program at least 6 times per week, and completed all outcomes at all time points.

ELIGIBILITY:
Inclusion Criteria:

* primary complaint of low back pain with or without leg symptoms
* duration of symptoms 24 hours to 90 days
* modified Oswestry score of 20 or greater
* able to read and speak English.

Exclusion Criteria:

* current pregnancy
* spinal steroid injections within the past month
* spinal surgery in the past 6 months
* current worker's compensation or motor vehicle accident claim
* presence of any red flag symptoms indicating possible serious pathology or non-musculoskeletal pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Modified Oswestry Disability Questionnaire (ODQ) score | Baseline, 4 weeks, 6 months
  A measure of self-reported disability with scores ranging from 0% to 100% disability.

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) score | Baseline, 4 weeks, 6 months
  An 11 point scale in which patients rate their pain numerically with "0" representing no pain and "10" representing excruciating pain.
Global Rating of Change (GRC) | 4 weeks, 6 months
  A self-report measure that asks subjects to rate the change in their symptoms from baseline. Scores range from +7 ("a very great deal better") to -7 ("a very great deal worse") with 0 representing no change.
Overall Treatment Success | 4 weeks, 6 months
  Success will be defined as a 50% or greater improvement in modified Oswestry Disability Questionnaire score, a decrease in Numeric Pain Rating Scale score of 3.5 points or greater, and Global Rating of Change score of +5 ("quite a bit better") or greater. If all three of these criteria are met, the overall outcome will be considered "successful". If one or more of these criteria is not met, overall outcome will be considered "unsuccessful".

OTHER OUTCOMES:
Total Number of Visits | At discharge, which will be approximately 4 weeks
  Total number of physical therapy visits completed.
Duration of Care | At discharge, which will be approximately 4 weeks
  The number of days from the first physical therapy visit to the last physical therapy visit.
Number of adverse events from treatment | up to 6 months
  Any adverse event reported as a result of treatment. Seriousness of adverse events will be graded on a 1 to 5 scale according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE) grading scale.
Number of patients seeking further treatment | 6 months
  Number of patients seeking further treatment (i.e. continued physical therapy, acupuncture, chiropractic treatment, spinal injections, or surgery) for their low back pain at 6 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: David W Candy, DPT, Principal Investigator — Hendricks Regional Health
Locations (1):
- Hendricks Regional Health, Plainfield, Indiana, United States

REFERENCES:
- [Background] Delitto A, Erhard RE, Bowling RW. A treatment-based classification approach to low back syndrome: identifying and staging patients for conservative treatment. Phys Ther. 1995 Jun;75(6):470-85; discussion 485-9. doi: 10.1093/ptj/75.6.470. PMID 7770494
- [Background] Fritz JM, Brennan GP, Clifford SN, Hunter SJ, Thackeray A. An examination of the reliability of a classification algorithm for subgrouping patients with low back pain. Spine (Phila Pa 1976). 2006 Jan 1;31(1):77-82. doi: 10.1097/01.brs.0000193898.14803.8a. PMID 16395181
- [Background] Fritz JM, Cleland JA, Childs JD. Subgrouping patients with low back pain: evolution of a classification approach to physical therapy. J Orthop Sports Phys Ther. 2007 Jun;37(6):290-302. doi: 10.2519/jospt.2007.2498. PMID 17612355
- [Background] Wainner RS, Whitman JM, Cleland JA, Flynn TW. Regional interdependence: a musculoskeletal examination model whose time has come. J Orthop Sports Phys Ther. 2007 Nov;37(11):658-60. doi: 10.2519/jospt.2007.0110. No abstract available. PMID 18057674
- [Background] Fritz JM, Delitto A, Erhard RE. Comparison of classification-based physical therapy with therapy based on clinical practice guidelines for patients with acute low back pain: a randomized clinical trial. Spine (Phila Pa 1976). 2003 Jul 1;28(13):1363-71; discussion 1372. doi: 10.1097/01.BRS.0000067115.61673.FF. PMID 12838091
- See also: Hendricks Regional Health — http://www.hendricks.org